CLINICAL TRIAL: NCT03483727
Title: Use of a Hand-held Digital Cognitive Aid in the Early Management of Simulated War
Brief Title: Use of a Hand-held Digital Cognitive Aid in the Early Management of Simulated War Wounds.
Acronym: SIMMAXMARCHE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Claude Bernard University (Other)
Responsible Party: Principal Investigator, CEJKA Jean-Christophe, MD, PhD, mEng, Claude Bernard University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ClaudeBernardU
Record Dates: First submitted 2018-03-23; First posted 2018-03-30 (Actual); Last update posted 2018-03-30 (Actual); Status verified 2018-03

CONDITIONS: Combat Casualty Care

STUDY DESIGN:
Intervention Model Description: with or without the cognitive aid
Who Masked: Participant
Masking Description: single
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digital cognitive aid (Experimental): The digital cognitive aid is designed as a smartphone app.
  Interventions: Device: SIMMAXMARCHERYAN
- no digital cognitive aid (Experimental): No cognitive aid in the hand of the leader during crises management.
  Interventions: Device: SIMMAXMARCHERYAN

INTERVENTIONS:
Device: SIMMAXMARCHERYAN — Digital cognitive aid during the management of simulated combat wounded.

SUMMARY:
Combat casualty care has proven to increase survival rate in military conflict by treating without delay the quickest-to-kill wounds. The French militaries are trained to the MARCHE RYAN acronym, an algorithm designed to help every soldiers provide simple treatment in order to bring the patient to the surgeon alive.

Our first study (MAX, Lelaidier et al, BJA 2017) clearly showed that the use of a digital cognitive aid in the hand of the leader significantly improves the management of anaesthesia & intensive care emergencies (malignant hyperthermia, anaphylactic shock, acute toxicity of local anaesthetics, severe and symptomatic hyperkalaemia).

The present study exclusively deals with the management of combat casualties with the same digital cognitive aid adapted for MARCHE RYAN algorithm.

DETAILED DESCRIPTION:
In a first study (MAX, BJA 2017, Lelaidier et al) the investigators designed a digital cognitive aid (MAX for Medical Assistant eXpert) under the form of a smartphone application including 5 scenarios of anaesthesia and intensive care crises (malignant hyperthermia, anaphylactic shock, acute toxicity of local anaesthetics, severe and symptomatic hyperkalaemia, ventricular fibrillation), designed to be used in the hand of the leader managing the situations. Technical and non-technical skills were improved in 4 out of 5 scenarios.

Combat casualties are dealt with a stereotyped management in the French army, and all soldiers learn the algorithm (acronym) designed for this purpose, the MARCHE RYAN. Situations requiring the use of the MARCHE RYAN are extremely stressful (on the battlefield, performed by non-medical personal, often on a comrade).

The present study exclusively deals with the management of combat casualties with the digital cognitive aid MAX adapted for MARCHE RYAN algorithm.

ELIGIBILITY:
Inclusion Criteria:

* Soldiers
* already trained in Combat Care level 2, under training for external operations.

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-05-31 (Actual); Study Completion 2017-09-01 (Actual)

PRIMARY OUTCOMES:
Technical Performance as compared to a Reference Task List | Time 0-30 min
  as compared to a Reference Task List

SECONDARY OUTCOMES:
Non technical skills performance | Time 0-30 min
  as measured by the Ottawa score

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Truchot M, Balanca B, Wey PF, Tazarourte K, Lecomte F, Le Goff A, Leigh-Smith S, Lehot JJ, Rimmele T, Cejka JC. Use of a Digital Cognitive Aid in the Early Management of Simulated War Wounds in a Combat Environment, a Randomized Trial. Mil Med. 2020 Aug 14;185(7-8):e1077-e1082. doi: 10.1093/milmed/usz482. PMID 32091610